CLINICAL TRIAL: NCT03010384
Title: Contact to a Physician Specialized in Social Medicine and the Impact on Return to Workforce in Patients Suspected of Disc Herniation? - a Randomized Controlled Trial
Brief Title: Contact to a Physician Specialized in Social Medicine and Return to Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsten Fonager (Other)
Responsible Party: Sponsor-Investigator, Kirsten Fonager, Consultant, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Reuma-2011
Record Dates: First submitted 2016-12-06; First posted 2017-01-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Return to Work; Musculoskeletal Disease
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): Consultation with a physician specialized in social medicine. The consultation lasted about one hour. Together with the patient a return-to-work (RTW) schedule was made to ascertain the need for contact to the workplace (to adjust work functions), municipality, general practitioner or short-term supportive consultations with a psychologist. If relevant, patients were offered up till 5 sessions with a psychologist.
  Interventions: Other: Rehabilitation program
- Control (No Intervention): Standard treatment from the Department of Rheumatology

INTERVENTIONS:
Other: Rehabilitation program
  Arms: Intervention

SUMMARY:
The aim of this study was to investigate the impact of a rehabilitation program including a physician specialized in social medicine parallel to treatment for suspected spinal disc herniation.

DETAILED DESCRIPTION:
In a two-year time period (2011 to 2012) 443 patients of suspected of disc herniation and risk of low work ability - based on questionnaires participated in a randomized control trial. The patients were randomized to either the intervention group (n=220) or control group (n=223). The intervention group were invited to the Department of Social Medicine two to four weeks after their first contact to Department of Rheumatology for a consultation with a physician specialized in social medicine. Together with the patient a return-to-work (RTW) schedule was made to ascertain the need for contact to the workplace (to adjust work functions), municipality, general practitioner or short-term supportive consultations with a psychologist. Throughout the intervention, the patients received their usual treatment from the Department of Rheumatology like patients from the control group. Outcome was return to the work force at one year follow up using information from a national registry.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 and < 60 years old,
* not receiving disability pension and not on maternity leave.
* sick leave over the past year for more than ten days
* low self-rated work ability for the next two years
* health anxiety

Exclusion Criteria:

-

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 443 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Return to Work (register based information) | one year